CLINICAL TRIAL: NCT04529863
Title: Data Analysis for Drug Repurposing for Effective Alzheimer's Medicines- Tocilizumab vs Abatacept
Brief Title: Data Analysis for Drug Repurposing for Effective Alzheimer's Medicines (DREAM) - Tocilizumab vs Abatacept
Acronym: DREAM
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Rutgers University (Other); Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Rishi J. Desai, Assistant Professor, Brigham and Women's Hospital
Other Study IDs: 2019A010961-1; 75N95019C00057 (Other Grant/Funding Number: National Institute on Aging)
Record Dates: First submitted 2020-08-25; First posted 2020-08-28 (Actual); Last update posted 2021-11-16 (Actual); Status verified 2021-11

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tocilizumab; Abatacept

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Tocilizumab: Reference group
  Interventions: Drug: Tocilizumab
- Abatacept: Exposure group
  Interventions: Drug: Abatacept

INTERVENTIONS:
Drug: Tocilizumab — Tocilizumab claim is used as the reference group.
  Groups: Tocilizumab
Drug: Abatacept — Abatacept claim is used as the exposure group.
  Groups: Abatacept

SUMMARY:
This study aims to evaluate the comparative risk of dementia/Alzheimer's disease onset between patients treated with medications that target specific metabolic pathways and patients treated with alternative medications for the same indication.

DETAILED DESCRIPTION:
This is a non-randomized, non-interventional study that is part of the DREAM Study of Brigham and Women's Hospital. DREAM is led by Dr. Madhav Thambisetty, MD, PhD, Chief of the Clinical and Translational Neuroscience Section, Laboratory of Behavioral Neuroscience, National Institute on Aging (NIA) intramural research program. This study aims to evaluate the comparative risk of dementia/Alzheimer's disease onset between patients treated with medications that target specific metabolic pathways and patients treated with alternative medications for the same indication using healthcare claims data.

ELIGIBILITY:
Please see https://docs.google.com/spreadsheets/d/1paz3s8atiPsH8kyaCgxB8gcqQYNnK1Cv_om79IfIAsI/edit?usp=sharing or Appendix A for full code and algorithm definitions.

Medicare timeframe: 2007 to 2017 (end of data availability).

Inclusion Criteria:

* 1. No prior use of tocilizumab or abatacept anytime prior to cohort entry date
* 2. Enrollment in Medicare Part A, B, and D with no HMO coverage for 365 days prior to and including cohort entry date

Exclusion Criteria:

* 1. Prior history of dementia measured anytime prior to cohort entry date
* 2. No prior history of rheumatoid arthritis recorded in the 365 days prior to cohort entry date
* 3. Prior history of nursing home admission in the 365 days prior to the cohort entry date

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will involve a new user, parallel group, cohort study design comparing tocilizumab to abatacept. The patients will be required to have continuous enrollment during the baseline period of 355 days before initiation of tocilizumab or abatacept (cohort entry date). Follow-up for the outcome (incident dementia), begins the day after drug initiation for analyses 1, 3, and 4 and 180 days after drug initiation for analysis 2.
Sampling Method: Non-Probability Sample
Enrollment: 30432 (Actual)
Dates: Start 2020-08-17 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Time to dementia onset | Through study completion (a median of 250 days)
  Time to dementia onset, i.e., Alzheimer's disease, vascular dementia, senile, presenile, or unspecified dementia, or dementia in other diseases classified elsewhere. Please refer to uploaded protocol for full definition due to size limitations.

SECONDARY OUTCOMES:
Time to Alzheimer's disease onset | Through study completion (a median of 250 days)
  Time to Alzheimer's disease onset. Please refer to uploaded protocol for full definition due to size limitations.

CONTACTS AND LOCATIONS:
Overall Officials: Rishi J Desai, PhD, Principal Investigator — Brigham and Women's Hospital; Madhav Thambisetty, MD, PhD, Principal Investigator — National Institute on Aging (NIA)
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-24): https://cdn.clinicaltrials.gov/large-docs/63/NCT04529863/Prot_SAP_003.pdf